CLINICAL TRIAL: NCT06891378
Title: Effects of Mobile App-based Self-rehabilitation for Patients After Reverse Total Shoulder Arthroplasty: Pilot Non-RCT
Brief Title: At Home, Digital Rehabilitation for Patients After Reverse Total Shoulder Arthroplasty
Acronym: DHI_RTSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-02-088; RS-2024-00401350 (Other Grant/Funding Number: Korea Health Industry Development Institute)
Record Dates: First submitted 2025-03-14; First posted 2025-03-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Arthroplasty, Replacement, Shoulder; Reverse Total Shoulder Arthroplasty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This non-randomized comparative study will prospectively recruit 30 participants to receive the intervention. Additionally, a retrospective cohort of approximately 70 patients will be selected using propensity score matching to serve as a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrevention group (mHealth group) (Experimental): The main characteristics of the intervention provided to the intervention group are as follows:
  1. Customized rehabilitation exercise program is assigned after surgery and rehabilitation exercise is performed while watching the video
  2. Recovery of shoulder joint range of motion can be checked through movement evaluation
  3. Exercise diary writing (exercise schedule and post-exercise condition can be checked)
  4. Activity amount can be checked through step count collection
  5. Exercise record is checked and, if exercise is not performed, reason is confirmed through contact
  Interventions: Other: Intrevention group (mHealth group)
- control group (usual care) (Active Comparator): This group performs home rehabilitation exercises using in-hospital educational materials. Control group data are retrospectively collected and matched using propensity score methods.
  Interventions: Other: control group (usual care)

INTERVENTIONS:
Other: Intrevention group (mHealth group) — 1. Receive a customized rehabilitation exercise program after surgery and perform rehabilitation exercises while watching videos
  2. Check recovery of shoulder joint range of motion
  3. Write an exercise diary (check exercise schedule and post-exercise condition)
  4. Check activity level through step count collection
  5. Check exercise records and contact to confirm reason if exercise was not performed
  Arms: Intrevention group (mHealth group)
Other: control group (usual care) — This group performs home rehabilitation exercises using in-hospital educational materials.
  Control group data are retrospectively collected and matched using propensity score methods.
  Arms: control group (usual care)

SUMMARY:
1. Why This Study Matters Over the past five years, more people in Korea have been having shoulder surgery. With our country moving into a super-aged society by 2025, these surgeries are expected to increase even more. More people today are focused on staying healthy and active, so many are choosing shoulder surgery to enjoy a better quality of life. According to the Health Insurance Review and Assessment Service, around 90,000 shoulder surgeries take place each year, and most of these patients (84.6%) are over 50.
2. Reverse Shoulder Arthroplasty (RTSA) and the Role of Rehabilitation RTSA is a type of shoulder surgery often used when there's extensive damage to the shoulder's rotator cuff. Its use is growing rapidly-making up about one-third of shoulder replacements in the United States and over 90% in some European countries. Although shoulder replacement surgeries are increasing worldwide, we still need more research on the best ways to help patients recover. In particular, we want to see if using a mobile app for self-guided rehabilitation can be effective.
3. The Need for Mobile App-Based Self-Rehabilitation After shoulder surgery, proper rehabilitation is crucial for a good recovery. Recent studies have shown that a mobile app can help patients easily follow their rehabilitation exercises. It also improves their understanding of the recovery process and keeps them more engaged in their treatment. Previous research has even shown that patients recovering from knee or hip replacement surgeries experienced better physical and mental recovery when using a mobile app.
4. Benefits of Using Technology for Rehabilitation Studies have found that patients who use remote rehabilitation techniques gain more confidence in managing their recovery on their own rather than relying solely on regular hospital visits. In one small study, five patients who used remote rehabilitation after RTSA reported high satisfaction with their recovery process. Mobile apps also allow healthcare providers to check that patients are doing their exercises correctly and to offer timely advice. This improved communication helps patients be more proactive about their recovery.
5. What This Study Aims to Do

This study will explore how mobile app-based self-rehabilitation affects recovery after shoulder replacement surgery. We will compare two groups of patients:

One group will use a mobile app to guide their rehabilitation. The other group will follow traditional rehabilitation instructions provided in a brochure.

ELIGIBILITY:
Inclusion criteria

* Those aged 50 or older
* Those who are indicated for and are scheduled to undergo reverse total shoulder arthroplasty (RTSA)
* Those who voluntarily decided to participate and gave written consent after hearing a detailed explanation of this study

Exclusion criteria

* Those who have difficulty using the application due to severe underlying diseases, neuromusculoskeletal diseases, cognitive or visual impairments, etc.
* Those with concomitant diseases such as neurological or visual impairments or uncontrolled cardiovascular disorders that make it difficult to participate in rehabilitation exercises
* Other people who, as determined by a medical professional, should not perform rehabilitation exercises without supervision

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the American Shoulder and Elbow Surgeons (ASES) Score from Preoperative Baseline to 12 Weeks | Before surgery, 12 weeks and 20 weeks after surgery
  It has a total range of 0 to 100 points (higher means better function). Pain is measured using the Visual Analog Scale (VAS, 10 points) and converted to 50 points, and function consists of 10 questions, each 0 to 3 points, a total of 30 points → converted to 50 points.

SECONDARY OUTCOMES:
Shoulder function - Korean shoulder score (KSS) | Before surgery, 12 weeks and 20 weeks after surgery
  The total score is 0-100 (the higher the better), and is composed of pain (30 points), function (40 points), activities of daily living (10 points), and muscle strength (20 points).
Shoulder function - Shoulder Simple Test (SST) | Before surgery, 12 weeks and 20 weeks after surgery
  The total score is 0 to 12 points (the higher the better the function), and there are 12 questions related to the function, with a yes/no response method. If you answer 'yes', you get 1 point, and the number of 'yes' answers is the total score.
Shoulder function - Constant Murley Shoulder Outcome Score | Before surgery, 12 weeks and 20 weeks after surgery
  Total 0~100 points (higher means better function), pain (15 points), activities of daily living (20 points), active joint range of motion (ROM) (40 points), muscle strength (25 points): Score is calculated by measuring strength in 90 degrees of abduction.
  In addition, an Adjusted Cnstant score will be calculated. This is adjusted for the Normal score (total 100 points) considering differences in shoulder function according to age and gender.
Pain - Visual Analog Scale (VAS) | Before surgery, 12 weeks and 20 weeks after surgery
  The higher the Visual Analog Scale (VAS, 0~10 points), the more pain there is.
Isokinetic Shoulder Mucle Strength | Before surgery, 12 weeks (only Isometric strength) and 20 weeks after surgery
  Isokinetic strength: Using an isokinetic strength measuring device called CSMi Medical Solutions, isokinetic strength (internal rotation, external rotation) for each movement is measured according to a standardized protocol. During the test, the subject is seated on a chair and the torso is fixed to the dynamometer. The subject is asked to hold the opposite handle of the dynamometer.
Active Shoulder range of moiton (degree) | Before surgery, 12 weeks and 20 weeks after surgery
  1. Flexion: Measure the maximum angle when the arm is raised forward according to the standard protocol.
  2. Abduction: Measure the maximum angle when the arm is raised sideways according to the standard protocol.
  3. External rotation: Collect the maximum angle measured when the arm is placed next to the trunk.
Shoulder range of moiton - internal rotation | Before surgery, 12 weeks and 20 weeks after surgery
  Internal rotation: Measure the position of the thumb tip on the spine level when the arm is sent behind the back. Each position is scored. (Thoracic T1-T12 = 1-12 points; Lumbar L1-L5 = 13-17 points; Hip = 18 points)
Passive Shoulder range of moiton (degree) | Before surgery, 12 weeks and 20 weeks after surgery
  1. Flexion: Measure the maximum angle when the arm is raised forward according to the standard protocol.
  2. Abduction: Measure the maximum angle when the arm is raised sideways according to the standard protocol.
  3. External rotation: Collect the maximum angle measured when the arm is placed next to the trunk.
Isometric Shoulder Mucle Strength | Before surgery, 12 weeks (only Isometric strength) and 20 weeks after surgery
  Using a hand-held dynamometer (FGN-20B, SHIMPO, JAPAN), the maximum force (in pounds) is collected and measured in the internal rotation (at side), external rotation (at side), and scaption positions.

OTHER OUTCOMES:
Self-efficacy for exercise (SEE) | Before surgery, 12 weeks and 20 weeks after surgery
  1. Consists of 9 items on situations that hinder exercise.
  2. Evaluate how confident you are that you can exercise 20 minutes 3 times a week in each situation on a scale of 10% intervals from 0% (not at all confident) to 100% (very confident).
  3. Interpret as '0-20% = not at all confident, 20-40% slightly confident, 40-60% = moderately confident, 60-80% = very confident, 80-100 = extremely confident.'
     * Collected only in prospective intervention group
EQ-5D-5L, Quality of Life | Before surgery, 12 weeks and 20 weeks after surgery
  The EQ-5D-5L is a standardized instrument developed by the EuroQol Group to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels. Index scores range from less than 0 (worse than death) to 1 (full health).
  This measure will be collected only in the prospective intervention group to evaluate changes in perceived quality of life during the rehabilitation process. Retrospective control data are not available for this outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Irwon-ro 81, South Korea

IPD SHARING:
Plan to Share IPD: No
Since this provides the subject's personal information to a third party, separate consent is required.